CLINICAL TRIAL: NCT05172427
Title: Acceptability/Feasibility Testing of an Intervention Targeting Intolerance of Uncertainty
Brief Title: Acceptability/Feasibility of IU Intervention
Acronym: CLUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor of Clinical Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BARLOW_CLUE intervention
Record Dates: First submitted 2021-09-08; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Generalized Anxiety Disorder; Emotional Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — elastin microfibril interface located protein

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two active conditions or a waitlist control condition. Participants assigned to the EMA/EMI condition will receive the intervention, following by two weeks of EMA with personalized EMI prompts sent to them based on their responses to the EMA questions. Participants assigned to the EMA condition will receive the intervention, followed by two weeks of EMA only (with no EMI prompts based on their responses). The waitlist control will not receive the intervention prior to completing two weeks of EMA, and will not receive EMI prompts based on their responses. Those in the waitlist control will be given the opportunity to receive the intervention at their one-month follow up appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CLUE intervention (EMA + EMI) (Active Comparator): Participants will complete baseline questionnaires, followed by seven days of baseline EMA. After seven days of baseline EMA, they will have a meeting with a clinician and be given the CLUE intervention targeting intolerance of uncertainty. Following this intervention, participants will be given 14 days of EMA, which will include EMI prompts that they come up with at the end of the CLUE intervention (framed as "key takeaways"). After the two week period of EMA/EMI, participants will complete a post-intervention questionnaires. In addition to similar questionnaires to those administered at baseline, acceptability and feasibility of the intervention will be assessed at post-intervention. One month after post-intervention, participants will complete a one-month follow up questionnaire battery, that will again ask about acceptability and feasibility of the intervention, as well as parallel questions from baseline and post-intervention.
  Interventions: Behavioral: 14 days of EMI; Behavioral: Uncertainty reappraisal training
- CLUE intervention (EMA only) (Active Comparator): Participants will complete baseline questionnaires, followed by seven days of baseline EMA. After seven days of baseline EMA, they will have a meeting with a clinician and be given the CLUE intervention targeting intolerance of uncertainty. Following this intervention, participants will be given 14 days of EMA. After the two week period of EMA, participants will complete a post-intervention questionnaires. In addition to similar questionnaires to those administered at baseline, acceptability and feasibility of the intervention will be assessed at post-intervention. One month after post-intervention, participants will complete a one-month follow up questionnaire battery, that will again ask about acceptability and feasibility of the intervention, as well as parallel questions from baseline and post-intervention.
  Interventions: Behavioral: Uncertainty reappraisal training
- Waitlist control (No Intervention): Participants will complete baseline questionnaires, followed by seven days of baseline EMA. After seven days of baseline EMA, participants will be assigned 14 days of EMA. After the two week period of EMA, participants will complete a post-intervention questionnaires. In addition to similar questionnaires to those administered at baseline. One month after the post-intervention questionnaires, participants will complete a one-month follow up questionnaire battery, that will include parallel questions from baseline and post-intervention. As these participants did not receive the intervention following their baseline EMA, they will be given the opportunity to schedule an appointment for the intervention after they have completed their one-month follow up questionnaire.

INTERVENTIONS:
Behavioral: 14 days of EMI — Following the intervention, participants will receive personalized prompts whenever they report elevated stress or anxiety. These prompts will be generated at the end of the intervention session, and will only be sent to individuals in the EMI condition.
  Arms: CLUE intervention (EMA + EMI)
Behavioral: Uncertainty reappraisal training — CLUE consists of an hour long intervention, followed by a 2-week long EMI. During the hour long intervention session, participants will receive psychoeducation (i.e., defining uncertainty), discuss myths associated with uncertainty (e.g., if I do not plan things, they will go poorly), and discuss behavioral experiments that can be done to challenge uncertainty beliefs.
  Arms: CLUE intervention (EMA + EMI); CLUE intervention (EMA only)

SUMMARY:
Anxiety disorders are prominent mental health burdens, affecting roughly 1 in 5 adults annually, and a third of individuals over the course of their life. These disorders are also impairing to individuals, with 23% of individuals with anxiety disorders describing their impairment as serious. Given the public health impact, it is crucial that interventions are designed to alleviate symptoms of anxiety, through reducing risk factors that predispose individuals to develop anxiety. One approach to do this is to develop brief interventions that could be administered virtually, which can then be supplemented using ecological momentary intervention (EMI) to reduce risk factors for anxiety disorders. In contrast to targeting more distant risk factors, targeting more direct risk factors, such as intolerance of uncertainty, could be used in the prevention and treatment of anxiety disorders.

DETAILED DESCRIPTION:
Anxiety disorders have been estimated to impact roughly 1 in 5 (19%) adults in the United States over the past year, and almost a third (31%) of adults in the United States over the course of their life. Further, these disorders are impairing to individuals; 23% of individuals with anxiety disorders describing their impairment as serious. Given this public health impact, it is crucial, that interventions are designed to alleviate symptoms of anxiety, or to reduce risk factors that may predispose individuals to develop anxiety. Further, it is expected that the COVID-19 will have long-lasting impacts on mental concerns worldwide. With these concerns come new opportunities to improve mental health care, through ultra-brief, self-paced, web-based interventions. These interventions are ideal to increase access to care given their high dissemination value and low cost. Building on prior experimental and intervention work conducted by Dr. Allan, we aim to conduct pilot testing of an ultra-brief, CBT-informed intervention targeting intolerance of uncertainty, or an extreme aversion to and fear of uncertainty.

Intolerance of uncertainty is an ideal construct to target in a broad web-based intervention given theoretical and empirical links between intolerance of uncertainty and a broad spectrum of anxiety and related disorders. Theoretically, intolerance of uncertainty amplifies the experience of stress and anxiety causing people to engage in maladaptive cognitive (e.g., worry) and behavioral (e.g., checking, avoidance) strategies to reduce distress, preventing an opportunity to habituate to the uncertainty. Empirically, a recent meta-analysis reported effect sizes (ds) ranging from .4 to .6 across generalized anxiety disorder, major depression, obsessive compulsive disorder, social anxiety disorder, panic disorder and agoraphobia, and eating disorders. Other studies have implicated intolerance of uncertainty in posttraumatic stress disorder as well as suicidal thought and behavior. More recent evidence has demonstrated that intolerance of uncertainty is not only a "fundamental fear" underlying anxiety disorder etiology but has also been implicated in a host of other mental health problems, including substance use. We recently examined the impact of intolerance of uncertainty on anxiety and depression during the COVID-19 pandemic over three months and found intolerance of uncertainty was concurrently associated with and significantly predictive of symptoms of generalized anxiety disorder and depression. Therefore, not only is there strong theoretical and empirical support for intolerance of uncertainty as a transdiagnostic risk factor for anxiety and related conditions, but there is also evidence that supports intolerance of uncertainty as particularly relevant to the current environmental conditions due to COVID-19.

To date, we have conducted the only pilot RCT of a CBT-based intervention (clinicaltrials.gov NCT04199884). In a sample of 84 participants with elevated intolerance of uncertainty during their screening appointment, we compared a researcher-facilitated Intolerance of Uncertainty Treatment (IUT) to a time-matched healthy living control condition. IUT contains psychoeducation, challenging negative automatic thoughts regarding uncertainty through "mythbusting" exercises, and designing behavioral experiments to challenge these negative automatic thoughts. In this study, significant, medium effect size differences (d = .46) emerged between IUT and the control condition, but not until the month 1 follow-up. In addition, reductions in intolerance of uncertainty served as indirect effects from treatment condition to anxiety and depression symptoms. Further, most people found the intervention easy to understand, helpful, and applicable to their daily lives. Building on this prior work, we plan to adapt the existing ultra-brief intolerance of uncertainty intervention to be disseminated via a web-based computerized platform. Given the flexibility afforded via this digital platform, we also propose to include ecological momentary intervention (EMI) to enhance learning through the application of critical interventions skills as needed. EMI is ideal for these brief interventions as it allows for participants to gain the much-needed practice of challenging negative automatic thoughts and completing behavioral experiments critical to internalizing the skills and strategies taught during the intervention. Similar augmentations to brief interventions for stress, generalized anxiety disorder, and panic disorder (d = .5) have been successful in enhancing intervention effects (i.e., an additional d of .4 to .6), further underscoring the promise of including EMI to optimize outcomes.

The goals specific to this project are to 1) engage stakeholders in the design of an ultra-brief intolerance of uncertainty intervention (Enhanced Intolerance of Uncertainty Treatment [E-IUT]) and 2) to conduct a pilot trial to evaluate the acceptability, feasibility, and preliminary effect size estimates of E-IUT, in support of a larger fully powered test of E-IUT.

ELIGIBILITY:
Inclusion Criteria:

* Elevated GAD symptoms (i.e., GAD-7 scores greater than or equal to 10)
* Elevated IU symptoms (i.e., IUS-12 scores greater than or equal to 28)
* Access to a device with internet connection

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 | One day after 14-day EMA/EMI
  The CSQ-8 is a 8-item self-report scale that assesses client satisfaction with a particular intervention/program. The CSQ-8 is completed by rating satisfaction with services on a 1-4 Likert-type scale
Client Satisfaction Questionnaire-8 | One month follow up
  The CSQ-8 is a 8-item self-report scale that assesses client satisfaction with a particular intervention/program. The CSQ-8 is completed by rating satisfaction with services on a 1-4 Likert-type scale
Feasibility of service | 14-day EMA/EMI
  Feasibility will also be determined based on response rates for EMA/EMI. If 80% of participants respond to 80% of the EMA prompts, this will be considered a feasible means of service delivery

SECONDARY OUTCOMES:
Intolerance of Uncertainty-12 | Baseline
  a 12-item scale for measuring trait IU. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future.
Intolerance of Uncertainty-12 | One day after 14-day EMA/EMI
  a 12-item scale for measuring trait IU. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future.
Intolerance of Uncertainty-12 | One month follow up
  a 12-item scale for measuring trait IU. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future.
PROMIS anxiety scale | Baseline
  The PROMIS Anxiety scale measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS anxiety scale | One day after 14-day EMA/EMI
  The PROMIS Anxiety scale measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS anxiety scale | One month follow up
  The PROMIS Anxiety scale measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS depression scale | Baseline
  The PROMIS Depression scale measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS depression scale | One day after 14-day EMA/EMI
  The PROMIS Depression scale measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS depression scale | One month follow up
  The PROMIS Depression scale measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS stress scale | Baseline
  The PROMIS Psychological Stress scale measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS stress scale | One day after 14-day EMA/EMI
  The PROMIS Psychological Stress scale measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always).
PROMIS stress scale | One month follow up
  The PROMIS Psychological Stress scale measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always).
Alcohol Use Disorder Identification Test (AUDIT) | Baseline
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior.
Alcohol Use Disorder Identification Test (AUDIT) | One day after 14-day EMA/EMI
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior.
Alcohol Use Disorder Identification Test (AUDIT) | One month follow up
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior.
Drug Use Disorders Identification Test (DUDIT) | Baseline
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior.
Drug Use Disorders Identification Test (DUDIT) | One day after 14-day EMA/EMI
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior.
Drug Use Disorders Identification Test (DUDIT) | One month follow up
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior.
COVID-19 impact battery short-form (CIB-SF) | Baseline
  A five item questionnaire designed by the investigators will be used to assess COVID-19 related worries and impairment.
COVID-19 impact battery short-form (CIB-SF) | One day after 14-day EMA/EMI
  A five item questionnaire designed by the investigators will be used to assess COVID-19 related worries and impairment.
COVID-19 impact battery short-form (CIB-SF) | One month follow up
  A five item questionnaire designed by the investigators will be used to assess COVID-19 related worries and impairment.
COVID-19 contraction questions | Baseline
  Participants will be asked if they have contracted COVID-19 and how severe their symptoms were.
COVID-19 contraction questions | One day after 14-day EMA/EMI
  Participants will be asked if they have contracted COVID-19 and how severe their symptoms were.
COVID-19 contraction questions | One month follow up
  Participants will be asked if they have contracted COVID-19 and how severe their symptoms were.
Insomnia Severity Index (ISI) | Baseline
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four, with higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Insomnia Severity Index (ISI) | One day after 14-day EMA/EMI
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four, with higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Insomnia Severity Index (ISI) | One month follow up
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four, with higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Penn State Worry Questionnaire (PSWQ) | Baseline
  The PSWQ is a 16-item measure used to measure the trait of worry. The process of worry is pervasive throughout all of the anxiety disorders (Barlow, 1988). The questionnaire correlates with many psychological measures related to worry and does not correlate with other measures more remote to the construct. Items are measured on a 5-point Likert-type scale ranging from Not at all typical of me (1) to Very typical of me (5).
Penn State Worry Questionnaire (PSWQ) | One day after 14-day EMA/EMI
  The PSWQ is a 16-item measure used to measure the trait of worry. The process of worry is pervasive throughout all of the anxiety disorders (Barlow, 1988). The questionnaire correlates with many psychological measures related to worry and does not correlate with other measures more remote to the construct. Items are measured on a 5-point Likert-type scale ranging from Not at all typical of me (1) to Very typical of me (5).
Penn State Worry Questionnaire (PSWQ) | One month follow up
  The PSWQ is a 16-item measure used to measure the trait of worry. The process of worry is pervasive throughout all of the anxiety disorders (Barlow, 1988). The questionnaire correlates with many psychological measures related to worry and does not correlate with other measures more remote to the construct. Items are measured on a 5-point Likert-type scale ranging from Not at all typical of me (1) to Very typical of me (5).
The Anxiety Depression Distress Inventory-27 (ADDI-27) | Baseline
  The ADDI-27 is a 27-item questionnaire that contains three empirically derived scales (Positive Affect, Somatic Anxiety, and General Distress), which are relevant dimensions of the tripartite model of affect. Items are measured on a 5-point Likert-type scale ranging from Not at all (1) to Extremely (5).
The Anxiety Depression Distress Inventory-27 (ADDI-27) | One day after 14-day EMA/EMI
  The ADDI-27 is a 27-item questionnaire that contains three empirically derived scales (Positive Affect, Somatic Anxiety, and General Distress), which are relevant dimensions of the tripartite model of affect. Items are measured on a 5-point Likert-type scale ranging from Not at all (1) to Extremely (5).
The Anxiety Depression Distress Inventory-27 (ADDI-27) | One month follow up
  The ADDI-27 is a 27-item questionnaire that contains three empirically derived scales (Positive Affect, Somatic Anxiety, and General Distress), which are relevant dimensions of the tripartite model of affect. Items are measured on a 5-point Likert-type scale ranging from Not at all (1) to Extremely (5).
Perseverative Thought Questionnaire (PTQ) | Baseline
  The PTQ is a 15-item measure of repetitive negative thinking (RNT). Perseverative thinking is repetitive, negative thoughts that persist intrusive to the point of being unproductive to the individual. The thought process and the individual seeing the thoughts as dysfunctional can also characterize this thinking. Items are measured on a 5-point Likert-type scale of Never (0) to Almost Always (4).
Perseverative Thought Questionnaire (PTQ) | One day after 14-day EMA/EMI
  The PTQ is a 15-item measure of repetitive negative thinking (RNT). Perseverative thinking is repetitive, negative thoughts that persist intrusive to the point of being unproductive to the individual. The thought process and the individual seeing the thoughts as dysfunctional can also characterize this thinking. Items are measured on a 5-point Likert-type scale of Never (0) to Almost Always (4).
Perseverative Thought Questionnaire (PTQ) | One month follow up
  The PTQ is a 15-item measure of repetitive negative thinking (RNT). Perseverative thinking is repetitive, negative thoughts that persist intrusive to the point of being unproductive to the individual. The thought process and the individual seeing the thoughts as dysfunctional can also characterize this thinking. Items are measured on a 5-point Likert-type scale of Never (0) to Almost Always (4).
Ruminative Response Scale (RRS) | Baseline
  The RRS includes 22 items describing responses to depressed mood that are focused on self (e.g., "I think back to other times I have been depressed"), focused on symptoms (e.g., "I think about how hard it is to concentrate"), or focused on the possible consequences and causes of their mood (e.g., "I go away by myself and think about why I feel this way").
Ruminative Response Scale (RRS) | One day after 14-day EMA/EMI
  The RRS includes 22 items describing responses to depressed mood that are focused on self (e.g., "I think back to other times I have been depressed"), focused on symptoms (e.g., "I think about how hard it is to concentrate"), or focused on the possible consequences and causes of their mood (e.g., "I go away by myself and think about why I feel this way").
Ruminative Response Scale (RRS) | One month follow up
  The RRS includes 22 items describing responses to depressed mood that are focused on self (e.g., "I think back to other times I have been depressed"), focused on symptoms (e.g., "I think about how hard it is to concentrate"), or focused on the possible consequences and causes of their mood (e.g., "I go away by myself and think about why I feel this way").
Positive and Negative Affect Schedule-SF | Baseline
  The PANAS SF scales with two higher order factors: positive affect and negative affect. The PANAS-SF consists of 20 words that describe different feelings and emotions. Participants will be asked to rate on a 5-point Likert-type scale of Very slightly or not at all (1) to Extremely (5) for the degree in which they feel each word.
Positive and Negative Affect Schedule-SF | One day after 14-day EMA/EMI
  The PANAS SF scales with two higher order factors: positive affect and negative affect. The PANAS-SF consists of 20 words that describe different feelings and emotions. Participants will be asked to rate on a 5-point Likert-type scale of Very slightly or not at all (1) to Extremely (5) for the degree in which they feel each word.
Positive and Negative Affect Schedule-SF | One month follow up
  The PANAS SF scales with two higher order factors: positive affect and negative affect. The PANAS-SF consists of 20 words that describe different feelings and emotions. Participants will be asked to rate on a 5-point Likert-type scale of Very slightly or not at all (1) to Extremely (5) for the degree in which they feel each word.
The Metacognition Questionnaire-30 (MCQ) | Baseline
  The MCQ s a 30-item self-report scale measuring beliefs about thinking (i.e., metacognitive beliefs), monitoring tendencies, and judgements considered to be the etiological basis of anxiety and depression within the metacognitive model of psychopathology. Each item is scored on a four-point Likert response scale ranging from 1 (do not agree) to 4 (agree very much),
The Metacognition Questionnaire-30 (MCQ) | One day after 14-day EMA/EMI
  The MCQ s a 30-item self-report scale measuring beliefs about thinking (i.e., metacognitive beliefs), monitoring tendencies, and judgements considered to be the etiological basis of anxiety and depression within the metacognitive model of psychopathology. Each item is scored on a four-point Likert response scale ranging from 1 (do not agree) to 4 (agree very much),
The Metacognition Questionnaire-30 (MCQ) | One month follow up
  The MCQ s a 30-item self-report scale measuring beliefs about thinking (i.e., metacognitive beliefs), monitoring tendencies, and judgements considered to be the etiological basis of anxiety and depression within the metacognitive model of psychopathology. Each item is scored on a four-point Likert response scale ranging from 1 (do not agree) to 4 (agree very much),
Firearm ownership | Baseline
  Participants will be given a brief 4-item questionnaire about firearm ownership.
Firearm ownership | One day after 14-day EMA/EMI
  Participants will be given a brief 4-item questionnaire about firearm ownership.
Firearm ownership | One month follow up
  Participants will be given a brief 4-item questionnaire about firearm ownership.
Oxford Covid-19 Vaccine Hesitancy Scale | Baseline
  The Oxford Covid-19 Vaccine Hesitancy Scale s seven-item measure that assesses hesitancy regarding the COVID-19 vaccine.
Oxford Covid-19 Vaccine Hesitancy Scale | One day after 14-day EMA/EMI
  The Oxford Covid-19 Vaccine Hesitancy Scale s seven-item measure that assesses hesitancy regarding the COVID-19 vaccine.
Oxford Covid-19 Vaccine Hesitancy Scale | One month follow up
  The Oxford Covid-19 Vaccine Hesitancy Scale s seven-item measure that assesses hesitancy regarding the COVID-19 vaccine.
EMA questions | 7-day EMA period
  EMA questions will be given 4 times per day in a 12 hour period. The first survey ("Morning survey") will be a survey that takes approximately 3 minutes to complete. The following surveys ("afternoon surveys") will take approximately a minute to complete. In the 14 day EMA/EMI period, those in the CLUE + EMI condition will receive intervention prompts based on their responses. For those in the CLUE and waitlist control condition, they will not receive intervention prompts based on their responses.
EMA questions | 14-day EMA/EMI period
  EMA questions will be given 4 times per day in a 12 hour period. The first survey ("Morning survey") will be a survey that takes approximately 3 minutes to complete. The following surveys ("afternoon surveys") will take approximately a minute to complete. In the 14 day EMA/EMI period, those in the CLUE + EMI condition will receive intervention prompts based on their responses. For those in the CLUE and waitlist control condition, they will not receive intervention prompts based on their responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvard Medical School, 2007. National Comorbidity Survey (NCS). (2017, August 21). Retrieved from https://www.hcp.med.harvard.edu/ncs/index.php. Data Table 2: 12-month prevalence DSM-IV/WMH-CIDI disorders by sex and cohort.
- [Background] Oglesby ME, Allan NP, Schmidt NB. Randomized control trial investigating the efficacy of a computer-based intolerance of uncertainty intervention. Behav Res Ther. 2017 Aug;95:50-57. doi: 10.1016/j.brat.2017.05.007. Epub 2017 May 11. PMID 28531873
- [Background] Shapiro, M. O., Allan, N. P., & Schmidt, N. B. (under review). A randomized control trial examining the efficacy of an intolerance of uncertainty focused psychoeducation intervention. 14.
- [Background] Boswell JF, Thompson-Hollands J, Farchione TJ, Barlow DH. Intolerance of uncertainty: a common factor in the treatment of emotional disorders. J Clin Psychol. 2013 Jun;69(6):630-45. doi: 10.1002/jclp.21965. Epub 2013 Feb 4. PMID 23381685
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Dugas MJ, Schwartz A, Francis K. Brief Report: Intolerance of Uncertainty, Worry, and Depression. Cognit Ther Res. 2004;28(6):835-842. doi:10.1007/s10608-004-0669-0
- [Background] Tolin DF, Abramowitz JS, Brigidi BD, Foa EB. Intolerance of uncertainty in obsessive-compulsive disorder. J Anxiety Disord. 2003;17(2):233-42. doi: 10.1016/s0887-6185(02)00182-2. PMID 12614665
- [Background] McEvoy PM, Hyett MP, Shihata S, Price JE, Strachan L. The impact of methodological and measurement factors on transdiagnostic associations with intolerance of uncertainty: A meta-analysis. Clin Psychol Rev. 2019 Nov;73:101778. doi: 10.1016/j.cpr.2019.101778. Epub 2019 Oct 31. PMID 31678816
- [Background] Raines AM, Oglesby ME, Walton JL, True G, Franklin CL. Intolerance of uncertainty and DSM-5 PTSD symptoms: Associations among a treatment seeking veteran sample. J Anxiety Disord. 2019 Mar;62:61-67. doi: 10.1016/j.janxdis.2018.12.002. Epub 2018 Dec 12. PMID 30572246
- [Background] Zerach G, Levi-Belz Y. Intolerance of Uncertainty Moderates the Association Between Potentially Morally Injurious Events and Suicide Ideation and Behavior Among Combat Veterans. J Trauma Stress. 2019 Jun;32(3):424-436. doi: 10.1002/jts.22366. Epub 2019 Feb 5. PMID 30720890
- [Background] Carleton RN. Fear of the unknown: One fear to rule them all? J Anxiety Disord. 2016 Jun;41:5-21. doi: 10.1016/j.janxdis.2016.03.011. Epub 2016 Mar 29. PMID 27067453
- [Background] Garami J, Haber P, Myers CE, Allen MT, Misiak B, Frydecka D, Moustafa AA. Intolerance of uncertainty in opioid dependency - Relationship with trait anxiety and impulsivity. PLoS One. 2017 Jul 31;12(7):e0181955. doi: 10.1371/journal.pone.0181955. eCollection 2017. PMID 28759635
- [Background] Grassi A, Gaggioli A, Behavior GR-C&, 2009 undefined. The green valley: the use of mobile narratives for reducing stress in commuters. liebertpub.com. https://www.liebertpub.com/doi/abs/10.1089/cpb.2008.0156?casa_token=byLouW-52ZcAAAAA:R7eHFRaJmuBay29q9Rzkhazn9jKeKZEpN_PDzWjAeM7GQRTWaSrV3M_EWPOhzsOO8S223f4JYmY. Accessed May 1, 2020.
- [Background] Kenardy JA, Dow MG, Johnston DW, Newman MG, Thomson A, Taylor CB. A comparison of delivery methods of cognitive-behavioral therapy for panic disorder: an international multicenter trial. J Consult Clin Psychol. 2003 Dec;71(6):1068-75. doi: 10.1037/0022-006X.71.6.1068. PMID 14622082
- [Background] Newman MG, Przeworski A, Consoli AJ, Taylor CB. A randomized controlled trial of ecological momentary intervention plus brief group therapy for generalized anxiety disorder. Psychotherapy (Chic). 2014 Jun;51(2):198-206. doi: 10.1037/a0032519. Epub 2013 Sep 23. PMID 24059730